CLINICAL TRIAL: NCT05972408
Title: Evaluation of Prevalence, Molecular and Genetic Backgrounds of Calcium-Based Stones Among Patients With Renal Calcular Disease in Mansoura Urology and Nephrology Center
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Abolazm, Lecturer, Mansoura University
Other Study IDs: MD.21.02.426
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Renal Calculi
Keywords: renal calculi, Renal Ca oxalate stones, VDR gene
MeSH Terms: conditions — Kidney Calculi | interventions — Receptors, Calcitriol; Receptors, Calcium-Sensing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: percutaneous nephrlolithotomy — Endoscopic removal of renal stones
Genetic: VDR gene, CASR gene — checking possible mutations of VDR and CASR genes

SUMMARY:
Evaluation of Prevalence, Molecular and Genetic Backgrounds of Calcium-Based stones among Patients with Renal Calcular Disease in Mansoura Urology and Nephrology Center

DETAILED DESCRIPTION:
Back ground: Nephrolithiasis is a prevalent disease with high morbidity, the incidence and prevalence of nephrolithiasis has risen worldwide. Calcium nephrolithiasis may be considered as a complex disease having multiple pathogenic mechanisms and characterized by various clinical manifestations. Both genetic and environmental factors may increase susceptibility to calcium stones. Polymorphisms of vitamin D receptor (VDR), calcium-sensing receptor gene (CASR) and AGXT have been associated with risk of urolithiasis, but, with inconsistent results and lack data from Egyptian population.

Objective: Therefore, the present study aims to investigate the prevalence, mutational profile for these genes in patients with Ca-based stones, admitted to Mansoura Urology and Nephrology Center.

Methodology: In this study, employing sequencing of the coding exons of the calcium-sensing receptor gene (CASR), vitamin D receptor (VDR) and AGXT for a 50 of Egyptian calcium kidney stone-formers and 20 control subjects. The results of the mutational profile data will be correlated with risk of stone recurrence over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients with unilateral or bilateral renal stones (de novo or recurrent) who were candidates for endoscopic or surgical intervention were included. Metabolic workup was done for selected patients with radio-opaque stones, while genetic testing was done for those with dominant Ca composition proven by postoperative stone analysis. Thirty healthy individuals with no urologic abnormalities were involved as control cases. Patients with renal calculi for whom metabolic and genetic testing were performed are designated "α" cases.

Exclusion Criteria:

* For metabolic and genetic testing, patients with a well-known lesion precipitating stone disease were excluded e.g. ureteric stricture, ureteropelvic or ureterovesical junction obstruction, urinary diversion, history of ureterovesical re-implantation as well as patients with non-Ca stones by post-operative stone analysis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with unilateral or bilateral renal stones (de novo or recurrent) who were candidates for endoscopic or surgical intervention
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
prevalence of Ca-based renal stones | two years
  Prevalence of Ca stones among patients with kidney stone disease admitted in Mansoura UNC throughout the study duration as assessed by infrared spectroscopic stone analysis
Genetic background of Ca based renal stones | two years
  Identification of metabolic derangement and genomic alterations in patients with renal Ca stones (CASR, and VDR genes)

SECONDARY OUTCOMES:
Stone recurrence | two years
  Evaluation of the possible correlation of detected genomic mutations assessed by genetic analysis with stone recurrence at 2 years following stone management.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Lu J, Lang Y, Liu T, Wang X, Zhao X, Shao L. Two novel AGXT mutations identified in primary hyperoxaluria type-1 and distinct morphological and structural difference in kidney stones. Sci Rep. 2016 Sep 20;6:33652. doi: 10.1038/srep33652. PMID 27644547